CLINICAL TRIAL: NCT06451653
Title: Effectiveness of Men in Maternity Health (MiM) Intervention on Male Involvement in Maternal Health Care to Improve Maternal Health Outcomes in Naypyitaw, Myanmar
Brief Title: Men in Maternity Health (MiM) in Myanmar
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Collaborators: Myanmar Health Network Organization (Other); Myanmar Maternal and Child Welfare Association (Unknown)
Responsible Party: Principal Investigator, May Chan Oo, Academic Researcher, Chulalongkorn University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CUCPHS-001
Record Dates: First submitted 2024-05-22; First posted 2024-06-11 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Maternal Health Care; Myanmar; Men in Maternity Health; Male Partner; Institutional Delivery
MeSH Terms: interventions — Menogaril; Methods

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Men in Maternity Health (MiM) Intervention (Experimental): The men in maternity health (MiM) education program provided male partners of pregnant women with comprehensive education on maternal health, covering topics such as pregnancy complications, obstetric danger signs, maternal health care (including antenatal, delivery, and postnatal care), the benefits of birth preparedness and complication readiness (BPCR), and safe delivery practices. Invitation letters were sent to male partners by public health supervisors every first and third week to encourage participation in the MiM program's activities, while maternal health education sessions were conducted every second and fourth week.
  Interventions: Behavioral: Men in Maternity Health (MiM) Intervention
- Control (No Intervention): Male partners in the control group can only receive routine maternal health education if they accompany their female partners to antenatal care services at health facilities.

INTERVENTIONS:
Behavioral: Men in Maternity Health (MiM) Intervention — The six-month MiM education program focused on maternal health education for male partners of pregnant women in the intervention area. Assigned midwives offered two-hour-long, face-to-face health education and discussion sessions at five selected health centres every second and fourth Sunday, respectively, to accommodate participants' work schedules. Attendance consistently remained high at 80% of participants every month, with home visits for absentees to provide health education.
  Arms: Men in Maternity Health (MiM) Intervention

SUMMARY:
World Health Organization integrated husband involvement into reproductive health programs to carry out safe motherhood successfully and therefore it has been encouraged as a new strategy to improve maternal health since 2000. In Myanmar, maternal health intervention and education programs for safe motherhood are progressing but maternal mortality is still high. Even though sufficient evidences prove that husband can influence maternal health care service utilization during pregnancy and there by positively impact obstetric emergency, few interventions have focused on husband directly to involve and also effectiveness of husband involvement intervention on birth preparedness and complication readiness for safe motherhood are still limited in Myanmar. Therefore, the objective of this study is to explore the effectiveness of the men in maternity health (MiM) intervention on male involvement in maternal health care, including its impact on knowledge about maternal health related issues, attitudes towards maternal health care and birth preparedness and complication readiness (BPCR) practices and improving institutional delivery rates for safe motherhood.

ELIGIBILITY:
Inclusion criteria:

For Men in Maternity health (MiM) Intervention; male partners who

* Aged ≥ 18 years
* Partners' pregnancies are ≤16 weeks gestational age
* Partners are pregnant for the first time (Gravida 1)
* Currently live with their female partners
* Have been living in the study area for at least 1 year

For quantitative and qualitative assessment:

* Male partners who participated in the MiM intervention and their female partners
* Maternal health stakeholders who oversee MiM implementation and maternal health care providers in the intervention township

Exclusion criteria:

For Men in Maternity Health (MiM) Intervention, male partners who

* Are severely ill and cannot communicate
* Do not give consent

For quantitative and qualitative assessment:

* Feel uncomfortable to participate in this study
* Do not give consent
* Are severely ill and cannot communicate

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2018-10-15 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Maternal Health Knowledge | 2 months pre-intervention and 2 months post-intervention
  To assess the effectiveness of the Men in Maternity Health (MiM) intervention on male involvement in maternal health, specifically regarding changes in maternal health knowledge, including knowledge of maternal health care, danger signs during pregnancy, delivery, and the postpartum period.
  Measurement: Pre- and post-intervention surveys assessed knowledge with 12 questions, each containing multiple sub-questions. Scoring was '1' for each correct answer, with a total score range from 0 to 36.
Attitudes Towards Maternal Health | 2 months pre-intervention and 2 months post-intervention
  To assess the effectiveness of the Men in Maternity Health (MiM) intervention on male involvement in maternal health, specifically regarding changes in attitudes towards maternal health.
  Measurement: Pre- and post-intervention surveys assessed attitudes with 12 questions. For positive statements, scores ranged from 4 (strongly agree) to 1 (strongly disagree), and for negative statements, scores ranged from 1 (strongly disagree) to 4 (strongly agree), with a total score range of 12 to 48.
Birth Preparedness and Complication Readiness (BPCR) Practices | 2 months pre-intervention and 2 months post-intervention
  The impact of the Men in Maternity Health (MiM) intervention on male involvement in birth preparedness and complication readiness (BPCR) practices was assessed through pre- and post-intervention surveys. BPCR practices include five key components: planning the health facility for birth, ensuring the presence of skilled birth attendants, arranging transportation for delivery or emergencies, identifying potential blood donors and saving money for delivery expenses. BPCR practices were measured with a composite score derived from responses to five components, each corresponding to one of the essential BPCR practices. Responses were scored '1' for 'Yes' and '0' for 'No'. The total BPCR score ranged from 0 to 5, with higher scores indicating better birth preparedness and complication readiness.
Acceptability and Feasibility of Men in Maternity Health (MiM) Intervention | Up to 2 months post-intervention
  To gain a comprehensive understanding of the impact of the MiM program, the acceptability and feasibility of the intervention were assessed through qualitative methods. This included semi-structured interviews with maternal health stakeholders engaged in the MiM program and focus group discussions with male participants who involved in the MiM program and their partners. Key areas explored included assessing the program's effectiveness in preventing maternal emergencies, promoting institutional deliveries and gathering participant satisfaction and feedback, and identifying the barriers and facilitators specific to the program's implementation. Data were analyzed using thematic analysis to identify themes and patterns related to the intervention's acceptability and feasibility of the intervention, highlighting common experiences, challenges and facilitators reported by participants and healthcare stakeholders, as well as identifying perceived benefits of the intervention.

SECONDARY OUTCOMES:
Institutional delivery | Up to 3 months post-intervention
  For institutional delivery outcomes, the place of delivery and the birth attendant for delivery were checked at the end of the study period through a post-intervention survey. The researcher validated the reported institutional deliveries by cross-referencing birth certificate records and obtaining information from the assigned area midwives.

CONTACTS AND LOCATIONS:
Overall Officials: May Chan Oo, Principal Investigator — College of Public Health Sciences, Chulalongkorn University, Bangkok, 10330, Thailand
Locations (1):
- Chulalongkorn University, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Undecided